CLINICAL TRIAL: NCT03405987
Title: Association of T1-mapping and LV Strain Analysis by CMR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Andreas Kammerlander, MD, Medical University of Vienna
Other Study IDs: T1-strain-2436
Record Dates: First submitted 2018-01-14; First posted 2018-01-23 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Myocardial Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECV < median
  Interventions: Diagnostic Test: Strain analysis by CMR
- ECV ≥ median
  Interventions: Diagnostic Test: Strain analysis by CMR

INTERVENTIONS:
Diagnostic Test: Strain analysis by CMR — Strain analysis by CMR will be performed

SUMMARY:
The association of T1-mapping (both native and ECV) and strain analysis of LV and RV by CMR will be assessed. Results from strain analysis will be investigated in terms of their prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* undergoing CMR
* willingness to participate

Exclusion Criteria:

* <18 years old
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing CMR for whatever reason will be invited to participate. A specific subgroup of patients are heart failure with preserved ejection fraction.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-07-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Association of native LV T1-values and strain analysis | Baseline
  Association of native LV T1-values and strain analysis by CMR
Association of ECV and strain analysis | Baseline
  Association of ECV and strain analysis by CMR
Association of strain analysis and outcome | 2 years
  Association of strain analysis by CMR and outcome (combination of cardiovascular hospitalization or death)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No